CLINICAL TRIAL: NCT05878678
Title: Prospective Phase II Randomized Clinical Study of the Accuracy of Multi-modal Guided Particle Radiotherapy for Postoperative Breast Cancer With Different Arm Position
Brief Title: Prospective Study of Particle Radiotherapy for Breast Cancer With Different Arm Position
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Qing Zhang,MD, Professor, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-Bca2022-03
Record Dates: First submitted 2023-04-30; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: immobilization positions; breast cancer; particle radiotherapy; dosimetry; multi-modal guided radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed positions of arm up (Active Comparator): Patients will receive particle radiotherapy in arm up position. Radiation: adjuvant hypofractionated intensity-modulated proton radiotherapy; For patients received modified radical mastectomy, Clinical Target Volume (CTV) 1: chest wall ± regional lymph drainage area, 40.05Gy (RBE) in 15 fractions with proton radiotherapy; For patients received lumpectomy, CTV1: whole breast ± regional lymph drainage area, 40.05 Gy (RBE) in 15 fractions with proton radiotherapy; CTVtb: tumor bed SIB（simultaneous integrated boost） to 48 Gy (RBE) in 15 fractions with proton radiotherapy.
  Interventions: Device: Fixed positions of arm down and arm up
- Fixed positions of arm down (Experimental): Patients will receive particle radiotherapy in arm down position. Radiation: adjuvant hypofractionated intensity-modulated proton radiotherapy; For patients received modified radical mastectomy, CTV1: chest wall ± regional lymph drainage area, 40.05Gy (RBE) in 15 fractions with proton radiotherapy; For patients received lumpectomy, CTV1: whole breast ± regional lymph drainage area, 40.05 Gy (RBE) in 15 fractions with proton radiotherapy; CTVtb: tumor bed SIB to 48 Gy (RBE) in 15 fractions with proton radiotherapy.
  Interventions: Device: Fixed positions of arm down and arm up

INTERVENTIONS:
Device: Fixed positions of arm down and arm up — In order to explore the accuracy of breast cancer patients' treatment positions and its impact on dose of the new fixation device in two different fixed positions of arm up and arm down, optimize the position fixed equipment and methods of particle radiotherapy for breast cancer, and then establish the precision process of particle radiotherapy for breast cancer under the guidance of multimodal images.

SUMMARY:
The optical body surface image (C-RAD) was used to guide and track the change of positions, and multimodal images (including 2D X-ray images, CT images and PET-CT images) were used to verify the treatment positions. In order to explore the accuracy of breast cancer patients' treatment positions and its impact on dose of the new fixation device in two different fixed positions of arm up and arm down, optimize the position fixed equipment and methods of particle radiotherapy for breast cancer, and then establish the precision process of particle radiotherapy for breast cancer under the guidance of multimodal images. In a word, this is a dosimetry and prospective Phase II randomized clinical study of the accuracy of multi-modal guided particle radiotherapy for postoperative breast cancer with different arm position.

DETAILED DESCRIPTION:
PET-CT: Positron Emission Tomography - Computed Tomography CT: Computed Tomography

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically (cytological or histological) confirmed breast cancer with positive lymph nodes and postoperative adjuvant radiotherapy
2. Exclude distant metastasis
3. No ipsilateral breast and breast radiation therapy
4. Exclude patients requiring axillary irradiation
5. Age 18-80 years old
6. General good health (Eastern Cooperative Oncology Group, ECOG 0-2)
7. No complications such as severe pulmonary hypertension, cardiovascular disease, peripheral vascular disease, or severe chronic heart disease that may affect radiotherapy.
8. Non-pregnant (confirmed by serum or urine β-HCG test) or lactating women
9. Patients must sign informed consent to receive radiotherapy.

Exclusion Criteria:

1. Pathology unapproved breast cancer
2. With distant metastasis
3. The ipsilateral breast or breast has received radiation therapy
4. Patients requiring axillary irradiation
5. The dose limit of organs at risk cannot reach the preset safe dose limit
6. Pregnancy (confirmed by serum or urine β-HCG test) or lactation
7. Poor general health, Karnofsky Performance Status (KPS)<70，or ECOG>2
8. Severe complications that may affect radiotherapy, including: a) Unstable angina pectoris, congestive heart failure, myocardial infarction requiring hospitalization in the past 6 months, b) acute bacterial or systemic fungal infection, c) hospitalization for exacerbations of chronic obstructive pulmonary disease (COPD) or other respiratory diseases
9. Unable to understand the purpose of treatment or unwilling to sign the treatment consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of multi-modal guided particle radiotherapy for postoperative breast cancer with different immobilization position | within 3 months after radiotherapy
  The optical body surface image (C-RAD) was used to guide and track the change of positions, and multimodal images (including 2D X-ray images, CT images and PET-CT images) were used to verify the treatment positions. In order to explore the accuracy of breast cancer patients' treatment positions and its impact on dose of the new fixation device in two different fixed positions of arm up and arm down, optimize the position fixed equipment and methods of particle radiotherapy for breast cancer, and then establish the precision process of particle radiotherapy for breast cancer under the guidance of multimodal images.

SECONDARY OUTCOMES:
Acute toxicities | within 3 months after radiotherapy
  Acute toxicities assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Late toxicities | > 3 months after radiotherapy
  Late toxicities assessed by Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European organization for research and treatment of cancer (EORTC)
Tumor local control rate | at 5 years post radiotherapy
Overall survival rate | at 5 years post radiotherapy
Progression free survival rate | at 5 years post radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China